CLINICAL TRIAL: NCT07189260
Title: Pre- and Postoperative Chest Therapy With Positive Expiratory Pressure (PEP) to Prevent Hospital-acquired Pneumonia in Patients Undergoing Hip Fracture Surgery
Brief Title: Pre- and Postoperative Chest Therapy With Positive Expiratory Pressure (PEP) to Prevent Hospital-acquired Pneumonia
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital Bispebjerg and Frederiksberg (Other)
Responsible Party: Principal Investigator, Charlotte Densing, Project nurse, University Hospital Bispebjerg and Frederiksberg
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: PEP trial
Record Dates: First submitted 2025-06-11; First posted 2025-09-23 (Actual); Last update posted 2025-09-23 (Actual); Status verified 2025-08

CONDITIONS: Hip Fractures (ICD-10 72.01-72.2)
Keywords: hip fracture; pneumonia; PEP therapy; positive expiratory pressure; RCT; hospital-acquired pneumonia; systematic treatment with PEP; osteoporosis; frailty; multimorbidity
MeSH Terms: conditions — Hip Fractures; Pneumonia; Healthcare-Associated Pneumonia; Osteoporosis; Frailty | interventions — Positive-Pressure Respiration

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Active (Active Comparator): Medical therapy device
  Interventions: Device: positive expiratory pressure
- Standard treatment (No Intervention): Standard treatment

INTERVENTIONS:
Device: positive expiratory pressure — PEP therapy
  Arms: Active

SUMMARY:
The goal of this clinical trial is to investigate whether pre- and postoperative treatment with systematic PEP therapy can prevent hospital-acquired pneumonia in patients with hip frac-ture. It will also learn about the barriers regarding PEP therapy in this group of patients.

* Does pre- and postoperative treatment with systematic PEP therapy prevent hospital-acquired pneumonia in patients with hip fracture?
* Which barriers do participants have regarding PEP therapy in this group of patients? Researchers will compare systematic PEP therapy to no intervention besides standard treat-ment to see if systematic therapy with PEP can prevent hospital-acquired pneumonia.

Participants will:

* Receive systematic PEP therapy during hospitalization or no intervention besides standard treatment
* Register the PEP therapy four times daily on a paper checklist. Failure to perform the treatment and the reason must also be documented on the checklist.

ELIGIBILITY:
Inclusion Criteria:

* Hip fracture regardless of age
* Cognitively well-functioning
* Able to understand the study and give informed consent
* Able to speak and understand Danish
* Resident of Region Hovedstaden or Region Sjælland

Exclusion Criteria:

* Cognitively impaired
* Unable to understand the study and give informed consent
* Pneumonia upon admission
* Delirium upon admission
* Pneumothorax

For patients with e.g. dementia or brain injury, the ability to give informed consent will be assessed individually.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 566 (Estimated)
Dates: Start 2024-02-19 (Actual); Primary Completion 2029-12-31 (Estimated); Study Completion 2030-12-31 (Estimated)

PRIMARY OUTCOMES:
The incidence of hospital-acquired pneumonia | During hospitalization, from intervention start to discharge, which is on average one week
  Primary Outcome is the incidence of hospital-acquired pneumonia in the control and intervention group. Documented in the Sundhedsplatformen and diagnosed with one ore more of the following:
  * Thoracic x-ray
  * Sputum culture
  * Auscultation
  * Infection markers

SECONDARY OUTCOMES:
Number of participants dead within 30-days after discharge | 30-day mortality, assessed 30 days after discharge from the orthopedic ward
  Number of participants dead within 30 days after discharge
Number of participants readmitted within 30-days after discharge | 30-day readmission post-discharge, assessed 30 days after discharge from the orthopedic ward
  Number of participants readmitted within 30 days after discharge
Incidence of delirium during hospitalization (journal entry, CAM-screening, diagnosis), up to 4 weeks. | During hospitalization, from intervention start to discharge, which is on average one week
  Incidence of delirium during hospitalization (journal entry, CAM-screening, diagnosis), up to 4 weeks.
Degree of regained basic mobility (Cumulated Ambulation Score - CAS) on the the day of discharge compared to the assement made at admission. | CAS the weeks up to hip fracture and CAS at discharge, which is on average one week after admission
  Degree of regained basic mobility (Cumulated Ambulation Score - CAS) on the the day of discharge compared to the assement made at admission. CAS values ranges from 0 to 6. A score of 6 represents an independant patient in regards to getting in and out of bed, sit-to-stand from a chair, and walking. A score of 0 represents a patient completely dependant on help getting in and out of bed, sit-to-stand from a chair, and walking.
Discharge destination (home, nursing home, care facility, rehab, another ward/hospital, etc.). Number of participants discharged to home, care facility, rehab, another hospital/ward or ot he discharge destination. | Assessed at discharge from the orthopedic department, which is on average one week efter admission
  Discharge destination (home, nursing home, care facility, rehab, another ward/hospital, etc.). Number of participants discharged to home, care facility, rehab, another hospital/ward or o the discharge destination.

CONTACTS AND LOCATIONS:
Locations (2):
- Denmark (2):
  - Bispebjerg & Frederiksberg Hospital, Copenhagen
  - Herlev & Gentofte Hospital, Herlev

IPD SHARING:
Plan to Share IPD: Yes
Access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), will be provided to anyone who wishes to access the data.
Supporting Information: Study Protocol, SAP